CLINICAL TRIAL: NCT00759239
Title: Phase IV Randomised Double-masked Clinical Trial: Assessing Morning Versus Evening Dosing of a Fixed Dose Combination of Travoprost 0.004% / Timolol Maleate 0.5% in Patients With Primary Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMD-06-02
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2012-01

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component), or ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): One drop of Travoprost 0.004% / Timolol maleate 0.5% in each eye at 9 am and 1 drop of Timolol vehicle as placebo in each eye at 9 pm for 12 weeks.
  Interventions: Drug: Travoprost 0.004% / Timolol maleate 0.5%
- 2 (Experimental): One drop of Timolol vehicle as placebo in each eye at 9 am and one drop of Travoprost 0.004% / Timolol maleate 0.5% in each eye at 9 pm for 12 weeks.
  Interventions: Drug: Travoprost 0.004% / Timolol maleate 0.5%

INTERVENTIONS:
Drug: Travoprost 0.004% / Timolol maleate 0.5% — Solution, morning dosing
  Arms: 1
Drug: Travoprost 0.004% / Timolol maleate 0.5% — Solution, evening dosing
  Arms: 2

SUMMARY:
The purpose of this study is to assess the IOP-lowering efficacy of a combination of Travoprost / Timolol maleate, dosed in the morning or in the evening, in patients with open-angle glaucoma or ocular hypertension, who have an insufficiently controlled IOP (mmHg), and are using prostaglandin analogue monotherapy.

ELIGIBILITY:
Inclusion:

* Male or female adult patients over the age of 18 years
* Current treatment with prostaglandin analogue monotherapy, IOP-lowering medication.
* Meet the following IOP entry criteria in at least one treated eye (mean IOP):

  * ≥ 19 mmHg
  * ≤ 28 mmHg
* The patient is willing and able to sign and date the Informed Consent Form. Patients who wear contact lenses will be able to participate in the study, provided that the contact lenses are removed before instillation of study medication, and that the patient agrees to wait a minimum of 15 minutes, before re-inserting the lenses.

Exclusion:

* Females of childbearing potential (i.e. - those who are not surgically sterilised at least three months prior to the study start, or are not at least one year post-menopausal), who are:

  * Currently pregnant
  * Have a positive result on a urine pregnancy test at the Eligibility Visit
  * Intend to become pregnant during the study period
  * Are breast-feeding
  * Are not using highly effective birth control measures, for example;
* Hormonal - oral, implanted, or injected contraceptives or;
* Mechanical - spermicide in conjunction with a barrier such a condom or diaphragm or;
* Intra-Uterine Device (IUD)
* Any form of glaucoma other than open-angle glaucoma (with or without a pigment dispersion or pseudo-exfoliation component).
* Current or previous therapy with another investigational agent, within 30 days prior to study entry.
* History of chronic or recurrent severe inflammatory eye disease (e.g., scleritis, uveitis, herpes keratitis), in either eye.
* History of ocular trauma within the past six months in either eye
* History of ocular infection or ocular inflammation within the past three months in either eye.
* History of clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment in either eye.
* History of any other severe ocular pathology (including severe dry eyes), in either eye that would preclude the administration of a topical prostaglandin analogue.
* Intraocular surgery within the past six months as determined by patient history and/or examination in either eye.
* Ocular laser surgery within the past three months as determined by patient history and/or examination in either eye.
* Any abnormality preventing reliable applanation tonometry of either eye.
* Angle grade less than Grade 2 in either eye, as measured by gonioscopy (extreme narrow angle with complete or partial closure), assessed within the previous 12 months.
* Cup/disc ratio greater than 0.80 in either eye, assessed within the previous six months.
* Severe central visual field loss in either eye, defined as a sensitivity of ≤ 10 bB in at least two of the four visual field test points, closest to the point of fixation, assessed within the previous six months.
* Unable to safely discontinue all IOP lowering medication, for a minimum period of 28 days prior to Baseline Visit.
* Unable to safely discontinue all glucocorticoid medications administered by any route. Before the Eligibility Visit, patients must have performed a Wash Out of at least four weeks for any intermittent glucocorticoid medications and must be able to remain off these medications for the duration of the study.
* Use of any additional topical or systemic ocular hyposensitive medication during the study.
* History of bronchial asthma, or severe chronic obstructive pulmonary disease that would preclude the safe administration of a topical beta-blocker.
* Less than 30 days stable dosing regimen before the Screening Visit of any non-glaucoma medications or substances administered by any route and used on a chronic basis that may affect IOP. These may include, but are not limited to the following:

  * Sympathomimetic agents
  * Antimuscarinic agents
  * Antihistamines
  * Phenothiazines
  * Tricyclic antidepressants
  * Beta-antagonist blocking agents
  * Alpha agonists
  * Alpha-adrenergic blocking agents
  * Calcium channel blockers
  * Angiotensin converting enzyme inhibitors
  * Cardiac gylcosides
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Reduction in intraocular pressure | week 4, week 12

SECONDARY OUTCOMES:
Adverse events | Week 4, week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Western Eye Hospital, London, United Kingdom

REFERENCES:
- See also: Results on European Database — https://www.clinicaltrialsregister.eu/ctr-search/search?query=EMD-06-02